CLINICAL TRIAL: NCT06584058
Title: [14C] A Single-center, Nonrandomized, Open, Single-dose Substance Balance Study of HPP737 in Healthy Subjects
Brief Title: HPP737 Substance Balance Study in Human
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Newsoara Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Newsoara HYK Biopharmaceutical (Shanghai) Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-HPP737-I-006
Record Dates: First submitted 2024-08-05; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All healthy subjects (Experimental)
  Interventions: Drug: HPP737

INTERVENTIONS:
Drug: HPP737 — [14C]HPP737 oral preparation, 20mg（150μCi）, once

SUMMARY:
Main research purpose

1. Quantitative analysis of the total amount of radioactivity in excreta (urine and feces) of male healthy subjects after oral administration of [14C]HPP737, to obtain the cumulative excretion rate and main excretion routes of human radioactivity;
2. To identify the main metabolites in the offspring of [14C]HPP737 in healthy male subjects, and to determine the main biotransformation pathway and main metabolite structure;
3. To investigate the distribution of total radioactivity in whole blood and plasma and the pharmacokinetics of total plasma radioactivity in healthy male subjects after a single oral administration of [14C]HPP737.

Participants will:

1. Take Investigational product once
2. Stay in the clinic about 7 days for checkups and tests
3. Report their symptoms

ELIGIBILITY:
Inclusion Criteria:

1. Chinese healthy adult males, aged 18-45 years (including boundary values);
2. The body weight of the subject is not less than 50kg, and the body mass index (BMI) is between 19.0 and 26.0kg/m2 (including the boundary value);
3. The subject has no sperm donation plan during the trial period and within six months after the completion of the trial, and the subject and his or her partner have no birth plan during the trial period and within six months after the completion of the trial and voluntarily take strict contraceptive measures (see Appendix 4 for details);
4. Fully understand the purpose and requirements of the trial, voluntarily participate in the clinical trial and sign the written informed consent, and be able to complete the whole process of the trial according to the requirements of the trial.

Exclusion Criteria:

1. Those who have undergone comprehensive physical examination, vital signs, laboratory examination (blood routine, blood biochemistry, coagulation test, urine routine, infectious disease screening, thyroid function, stool routine + occult blood), chest X-ray (positive position), anal digital examination, abdominal B-ultrasound (liver, bile, pancreas, spleen and kidney), urinary system B-ultrasound, and heart color ultrasound with clinical significance;
2. During the screening period, any ECG abnormalities determined by the investigators to be clinically significant, including but not limited to electrocardiograms with machine reading abnormalities: Fridericia's formula (QTcF=QT/ (RR^0.33)) corrected QT interval (QTcF) >450 msec, QRS>110 msec, frequent atrial or ventricular premature beats;
3. Patients with abnormal color vision, retinitis pigmentosa, macular degeneration, nonarteriotic anterior ischemic optic neuropathy (NAION), or other fundus history deemed unsuitable by the investigators;
4. Allergic constitution, such as people who are known to be allergic to two or more substances, or have allergic diseases, or have a history of allergy to PDE4 inhibitors or similar drugs or their excipients;
5. Habitual constipation or diarrhea, a history of malabsorption syndrome, or a history of severe nausea, vomiting, diarrhea, and constipation within one week before the screening period;
6. have difficulty swallowing or any condition that may affect drug absorption (e.g., gastrectomy, cholecystectomy, gastric bypass, duodenotomy, colectomy);
7. Have a history of clinically serious disease or any disease or condition that the investigator believes may affect the test results, including but not limited to a history of digestive, circulatory, respiratory, endocrine, nervous, urinary, or blood, immune, psychiatric, or metabolic diseases;
8. Previous history of organic heart disease, heart failure, myocardial infarction, angina pectoris, torsional ventricular tachycardia, ventricular tachycardia, QT prolongation syndrome or family history (genetic proof or close relatives at a young age due to sudden cardiac death);
9. Major surgery or surgical incision not fully healed within 6 months prior to screening; Major surgery includes, but is not limited to, any surgery where there is a significant risk of bleeding, extended period of general anesthesia, or open biopsy or significant traumatic injury;
10. Previous active bleeding (such as peptic ulcer, intracranial hemorrhage, skin ecchymosis, gingival bleeding); History of any medical condition that may increase the risk of bleeding (e.g. tumor bleeding, spontaneous hematoma, eye bleeding, hemoptysis, gastrointestinal bleeding or ulcers, hematuria, reproductive system bleeding, traumatic hematoma/bleeding and recurrent epistaxis/gingival bleeding/subcutaneous or skin bleeding, etc.) within 6 months prior to screening;
11. Hemorrhoids or perianal disease accompanied by regular/blood in the stool, or positive stool occult blood test during the screening period;
12. Use of any drug that affects drug metabolism enzymes or transporters (P-gp and BCRP) in the 30 days prior to screening, as detailed in Appendix 5;
13. Have taken any prescription drugs, over-the-counter drugs, Chinese herbs or food supplements (vitamins, calcium supplements) in the 14 days prior to screening and before dosing;
14. Those who have taken any clinical trial drug or participated in any other clinical trial (including drug and device clinical trials) within 3 months prior to the screening period;
15. Those who have lost blood or donated blood (≥400mL) within 3 months before screening, or received blood transfusion or blood components within 1 month, or plan to donate blood within 3 months after the end of this trial;
16. Smokers who smoked more than 5 cigarettes per day or habitually used nicotine-containing products in the 3 months prior to the screening period, or were unable to stop using any tobacco products during the trial period;
17. Regular alcohol consumption in the six months prior to screening, i.e. drinking more than 14 units of alcohol per week (1 unit =285mL of beer or 25mL of 40% alcohol spirits or 100mL of wine), or a positive alcohol breath test, or unable to abstain during the test period;
18. Drug abuse or drug use history, or drug abuse screening positive;
19. Habitual or excessive (more than 8 cups a day, 1 cup =250mL) consumption of grapefruit juice, tea, coffee and/or caffeinated beverages, and unable to abstain during the trial period;
20. Those who have special requirements for diet and cannot comply with a unified diet;
21. Workers who require long-term exposure to radiation, or who have had significant radiation exposure (≥2 chest/abdominal CT, or ≥3 other types of X-rays) in the year prior to administration, or who have participated in radiopharma labeling tests;
22. Patients with a history of needle fainting and blood fainting, difficulty in blood collection or inability to tolerate venous puncture blood collection;
23. Those who had been vaccinated within 1 month prior to screening or planned to be vaccinated during the trial period;
24. Subjects whose compliance is considered poor by the investigator, or who have other factors unsuitable for participation in this trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Cmax (peak concentration) | Up to 12 months
  radiation pharmacokinetic parameter
Tmax (peak time) | Up to 12 months
  radiation pharmacokinetic parameter
AUC0-T (area under drug time curve) | Up to 12 months
  radiation pharmacokinetic parameter
AUC0-∞ (area under drug time curve) | Up to 12 months
  radiation pharmacokinetic parameter
t1/2 (elimination half-life) | Up to 12 months
  radiation pharmacokinetic parameter
CL/F (apparent clearance) | Up to 12 months
  radiation pharmacokinetic parameter
Vd/F (apparent volume of distribution) | Up to 12 months
  radiation pharmacokinetic parameter
MRT (mean residence time) | Up to 12 months
  radiation pharmacokinetic parameter
Cumulative drug excretion(Urine) | Up to 12 months
  Radioactive excretion corresponding to urine samples
Cumulative drug excretion(stool) | Up to 12 months
  Radioactive excretion corresponding to stool samples
Major metabolite | Up to 12 months
  The main metabolites in plasma, urine and fecal samples were identified by liquid chromatography-mass spectrometry (LC-MS), and radioisotope metabolites were analyzed to provide the main biotransformation pathway of HPP737 in human body.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Pan, Master, Principal Investigator — Second Affiliated Hospital of Soochow University
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided